CLINICAL TRIAL: NCT02827279
Title: Study of the Strategies of Visual Perception of Social Scenes During Emotional States Induced to Subjects With an Intrusive Disorder of the Development: Pilot Study
Brief Title: Study of the Visual Perception During Emotional States on Subjects With an Intrusive Disorder of the Development
Acronym: VisioTED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of inclusion period
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8991
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Emotion
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Other): Mesure of emotional induction by eye tracking on Patient with Pervasive Developmental Disorders (PDD)
  Interventions: Other: emotional induction
- Healthy volunteers (Other): Mesure of emotional induction by eye tracking on People without disorders
  Interventions: Other: emotional induction

INTERVENTIONS:
Other: emotional induction — The eye-tracking mesure the reaction at emotional induction using of sound stimuli in a group of children with or without ASD, in a context of

SUMMARY:
The Pervasive Developmental Disorders (PDD) are severe neurodevelopmental disorders, affecting nearly 1% of the general population. The disorder of social interaction has often been described as resulting from poor emotion recognition, or a bad perception of biological motion. However, the results of studies on these issues are very divergent. The PDD also been described as a disorder of emotion regulation, but few studies address the emotional feelings of individuals with ASD and their neuropsychological implications.

The main objective is to study the effect of induced emotion in the children with ASD on his visual exploration strategies.

This is a comparative exploratory pilot study. We'll look at using the eye-tracking, policy terms of the look in a group of children with ASD, in a context of emotional induction (joy, fear, sadness or anger) using of sound stimuli.

DETAILED DESCRIPTION:
Context: The Pervasive Developmental Disorders (PDD) are severe neurodevelopmental disorders, affecting nearly 1% of the general population. The disorder of social interaction has often been described as resulting from poor emotion recognition, or a bad perception of biological motion. However, the results of studies on these issues are very divergent. The PDD also been described as a disorder of emotion regulation, but few studies address the emotional feelings of individuals with ASD and their neuropsychological implications. Many studies analyzing the effect of emotions induced - or felt - in healthy subjects. The effect of emotion on cognitive or attentional process is often called "emotional effect of interference." As has already been demonstrated, an emotion (eg induced by music or film) results in a change in visual perception of the environment strategies. These non-conscious mechanisms promote interactive synchrony with the surrounding world, especially during social interactions. We then assumed that the alteration of these perceptual-emotional regulation processes in PDD contribute to disorders of social interactions. In the absence of sufficient data in the literature, we wish to establish an exploratory study using the Eye-tracking, to objectify the links between emotional and perceptual processing in PDD.

Objectives: The main objective is to study the effect of induced emotion in the children with ASD on his visual exploration strategies. We assume that the direction of gaze to photographs of different emotional valences in individuals with ASD is not changed by the emotional state in which they are located. We will compare a population of children with PDD in a control population matched for age, sex. Our secondary goal is to study the link between 1) the socio adaptive level (measured by the Vineland 2) the intensity of autistic symptoms (score ADI) and gaze orientation towards social subjects with visual stimuli.

Methods: This is a comparative exploratory pilot study. We'll look at using the eye-tracking, policy terms of the look in a group of children with ASD, in a context of emotional induction (joy, fear, sadness or anger) using of sound stimuli.

Conclusion: This study would better characterize the emotional processing in ASD and generate hypotheses that could be tested in other neurophysiological studies. Moreover, it can contribute to the development of new supported techniques.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Asperger syndrome or infantile autism (F84.0 et F84.5, classification CIM10, 1992).
* Total score in the algorithm of ADI and ADOS > at the threshold required for the diagnosis of disorders(confusions) of the autistic spectre
* Intelligence quotient verbal (IQ) upper to 70 in the various tests psychométriques
* Chronological age from 8 to 12 years
* Written consent signed by the parents and the child
* Affiliation or recipient with the mode of social security.

Exclusion Criteria:

* Consent refusal of the child or parents
* Presence of neurovisual disorder

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Ratio corresponding to the relative change in visual orientation | 1 hour
  mesured by eye tracking before and after each emotional induction

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Henry, MD, Principal Investigator — CHU de Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No